CLINICAL TRIAL: NCT06875791
Title: A Safety and Efficacy Trial of TV5M01 for Radiation-Induced Mucositis in Patients Undergoing Treatment for Head and Neck Cancer
Brief Title: Safety and Efficacy Trial of TV5M01 for Radiation-Induced Mucositis in Head and Neck Cancer Patients.
Acronym: TEMOR
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Principal Investigator, Angela Zambrano, Principal Investigator, Fundacion Clinica Valle del Lili
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025.18; 2025.18 (Other: Hospital Universitario Valle del Lili)
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Oral Mucositis
Keywords: Oral mucositis; Squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Stomatitis; Carcinoma, Squamous Cell | interventions — Tea; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TV5M01 Oral Gel for Radiation-Induced Mucositis (Experimental): This arm will receive TV5M01 oral gel (5% green tea extract with 0.1% morphine) as an oral rinse. Participants will use 10 mL of the preparation three times daily at 8-hour intervals (±2 hours) from the diagnosis of grade 1 or higher mucositis throughout radiation therapy or until mucositis resolves. The medication should be administered at consistent times daily without fasting requirements. Doses vomited while in clinic may be replaced; however, participants should not take replacement doses for self-administered doses vomited at home. Missed doses should be skipped rather than doubled at the next scheduled time.
  Interventions: Combination Product: Green Tea Extract with Morphine
- Triple Mixture Oral Rinse for Radiation-Induced Mucositis (Active Comparator): This arm will receive a Triple Mixture oral rinse (combination of 0.19% w/w Lidocaine, 0.29% w/w Nystatin, and 5.50% w/v Hydroxides). Participants will use 10 mL of the preparation three times daily at 8-hour intervals (±2 hours) from the diagnosis of grade 1 or higher mucositis until mucositis resolves. The medication should be administered at consistent times daily without fasting requirements. Doses vomited while in clinic may be replaced; however, participants should not take replacement doses for self-administered doses vomited at home. Missed doses should be skipped rather than doubled at the next scheduled time.
  Interventions: Combination Product: Active Comparator: Triple Mixture Oral Rinse for Radiation-Induced Mucositis

INTERVENTIONS:
Combination Product: Green Tea Extract with Morphine — TV5M01 is a novel oral rinse combining 5% green tea extract with 0.1% morphine in a gel formulation specifically designed for the treatment of radiation-induced oral mucositis. This unique combination leverages the antioxidant and anti-inflammatory properties of green tea polyphenols (particularly EGCG) with the analgesic effects of morphine delivered directly to the oral mucosa. Unlike other interventions, this formulation is administered as a 10 mL rinse three times daily with subsequent ingestion, targeting both local tissue healing and pain relief through a dual-action mechanism.
  Arms: TV5M01 Oral Gel for Radiation-Induced Mucositis
Combination Product: Active Comparator: Triple Mixture Oral Rinse for Radiation-Induced Mucositis — This arm will receive a Triple Mixture oral rinse (combination of 0.19% w/w Lidocaine, 0.29% w/w Nystatin, and 5.50% w/v Hydroxides). Participants will use 10 mL of the preparation three times daily at 8-hour intervals (±2 hours) from the diagnosis of grade 1 or higher mucositis until mucositis resolves. The medication should be administered at consistent times daily without fasting requirements. Doses vomited while in clinic may be replaced; however, participants should not take replacement doses for self-administered doses vomited at home. Missed doses should be skipped rather than doubled at the next scheduled time
  Arms: Triple Mixture Oral Rinse for Radiation-Induced Mucositis

SUMMARY:
This study is a Phase 2, double-blind, randomized controlled trial evaluating the safety and efficacy of TV5M01 (a 5% green tea and 0.1% morphine gel) compared to triple mixture (0.19% lidocaine, 0.29% nystatin, and 5.50% hydroxides) for treating radiation-induced oral mucositis in patients with head and neck squamous cell carcinoma.

The trial will enroll 40 patients (20 per group) with stage III-IV head and neck cancer receiving radiotherapy who develop grade 1 or higher mucositis. Participants will apply the assigned mouthwash three times daily from mucositis diagnosis until resolution.

Primary outcomes include safety (incidence of infections and adverse events) and efficacy (duration of grade 3-4 mucositis, days with severe pain). Secondary outcomes include quality of life and analgesic use. Randomization will use minimization methodology to balance important prognostic factors.

The study design incorporates two interim analyses after 10 and 19 participants, with clear safety monitoring and stopping rules. If successful, this trial could provide an evidence-based treatment option for radiotherapy-induced mucositis, potentially improving treatment completion rates and quality of life for head and neck cancer patients.

DETAILED DESCRIPTION:
Detailed Description

This Phase 2a randomized, double-blind controlled trial evaluates the efficacy and safety of TV5M01 (a 5% green tea extract and 0.1% morphine gel) for treatment of radiation-induced oral mucositis in head and neck cancer patients. Mucositis affects virtually all patients receiving radiotherapy for head and neck cancer, causing significant pain, impaired nutrition, and often necessitating treatment interruptions. Despite its prevalence, no effective evidence-based treatments exist.

The scientific rationale for TV5M01 combines two complementary mechanisms: the antioxidant and anti-inflammatory properties of green tea extract (epigallocatechin gallate) and the targeted analgesic effects of low-dose morphine. Preclinical studies demonstrate that EGCG inhibits radiation-induced cellular damage through multiple pathways, including reduction of reactive oxygen species, attenuation of pro-inflammatory cytokine expression, and mitigation of DNA damage. Topical morphine provides localized pain relief with minimal systemic absorption through peripheral opioid receptors that become upregulated in inflamed tissues.

This single-center trial will enroll 40 participants with stage III-IV squamous cell carcinoma of the head and neck who develop grade 1 or higher mucositis during radiotherapy. Participants will be randomized in a 1:1 ratio to receive either TV5M01 or triple mixture ("magic mouthwash" containing lidocaine, nystatin, and hydroxides) as 10mL oral rinses administered three times daily until mucositis resolution. The randomization employs a minimization algorithm to balance treatment groups across key prognostic factors including age, sex, tumor location, and histopathological grade.

To maintain blinding, both preparations will appear similar and will be dispensed in identical amber PET bottles. Stability studies confirm a 7-day shelf life when stored at 5°C. Comprehensive assessments include daily mucositis grading, pain scores, weekly oropharyngeal examinations with photographic documentation, and quality of life measures.

The trial incorporates robust safety monitoring with two planned interim analyses (after 13 and 26 participants). An independent Safety Monitoring Committee will review all adverse events and has authority to recommend early termination if safety concerns arise. Statistical analysis will employ non-parametric methods for efficacy comparisons, with sensitivity analyses using exact permutation techniques.

If successful, this trial could establish TV5M01 as an evidence-based treatment for radiation-induced mucositis, potentially improving treatment adherence and quality of life for head and neck cancer patients. The dual mechanism targeting both inflammation and pain represents an innovative approach to this challenging clinical problem that has remained largely unsolved despite decades of research.

A

y los subtitulos de imporancia Detailed Description Background and Significance

Head and neck squamous cell carcinoma represents a significant global health burden with increasing incidence in low and middle-income countries. Radiotherapy remains a cornerstone treatment modality, but oral mucositis develops in virtually 100% of patients receiving radiotherapy to the head and neck region. This complication frequently necessitates treatment modifications, potentially compromising oncologic outcomes and substantially impairing quality of life.

Despite its prevalence and clinical impact, current treatment options for radiation-induced mucositis remain suboptimal. The commonly used "magic mouthwash" preparations have demonstrated limited efficacy in controlled trials and face challenges with coverage of affected areas and patient-reported adverse effects.

Scientific Rationale

The TV5M01 formulation combines two active components with complementary mechanisms targeting the pathophysiology of radiation-induced mucositis:

The green tea extract (5%) contains epigallocatechin gallate (EGCG), which possesses potent antioxidant properties. In preclinical models, EGCG has demonstrated ability to inhibit radiation-induced apoptosis, reduce reactive oxygen species production, and attenuate pro-inflammatory pathways through NF-κB modulation.

The morphine component (0.1%) provides targeted analgesia through peripheral opioid receptors that become upregulated in inflamed tissues. The pharmacokinetic profile supports limited systemic absorption when applied topically, providing site-specific pain relief without significant central effects.

Study Design and Methodology

This trial employs a randomized, double-blind, controlled, parallel-group design to evaluate the superiority of TV5M01 compared to triple mixture. The study will enroll 40 participants allocated in a 1:1 ratio to either intervention or control groups.

Both preparations will be administered as 10mL oral rinses three times daily at 8-hour intervals, beginning upon diagnosis of grade 1 or higher mucositis and continuing until resolution or completion of radiotherapy.

Randomization and Blinding

The study utilizes a minimization randomization algorithm implemented through the REDCap platform to ensure balanced treatment groups across key prognostic factors including sex, age, tumor location, and histopathological grade.

To maintain blinding, both preparations will appear similar in color and consistency, will be dispensed in identical amber PET bottles, and will be labeled with participant identification codes only.

Monitoring and Safety Provisions

An independent Safety Monitoring Committee will oversee trial conduct and participant safety. Two formal interim analyses are planned after enrollment of 13 and 26 participants, respectively.

Pre-specified stopping rules include development of severe adverse events causally related to TV5M01, evidence of significant treatment inferiority at interim analyses, and regulatory safety alerts involving study components.

Anticipated Impact

If TV5M01 demonstrates superior efficacy compared to current standard approaches, it could significantly improve the management of radiation-induced mucositis, potentially enabling better adherence to planned radiotherapy regimens and enhancing quality of life during treatment. The dual-mechanism approach targeting both inflammatory processes and nociception represents an innovative strategy in addressing this challenging complication.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years and < 60 years

Diagnosis of HNSCC of the oral cavity, larynx, oro- and hypopharynx, diagnostic stage III-IV according to the AJCC 8th edition, scheduled to start radiotherapy

Ability to swallow solids and liquids before starting radiotherapy treatment

Adequate contraception for both sexes:

For women: negative pregnancy test for women of childbearing age; must be surgically sterile, postmenopausal (defined as absence of menstrual cycle for at least 12 consecutive months), or comply with an acceptable contraceptive regimen during and 3 months after the treatment period

For men: must be surgically sterile or comply with a contraceptive regimen during and for 3 months after the treatment period

Performance status (ECOG) of 0-1, measured within 72 hours prior to treatment initiation

Expected life expectancy ≥ 6 months

Adequate renal function [creatinine ≤ 1.5 times the upper limit of normal (ULN) or Glomerular Filtration Rate ≥ 50 ml/min]

Adequate liver function [total bilirubin ≤ 1.5 x ULN; AST or ALT ≤ 3 x ULN or ≤ 5 x ULN if due to tumor liver involvement]

Provision of signed and dated informed consent before initiating any study-related procedure

Meeting the diagnostic criteria for grade 1 or higher mucositis according to WHO classification

Meeting the criteria for starting radiotherapy

Willing and able to participate in the trial and comply with all trial requirements

Exclusion Criteria:

Patients not eligible for radiotherapy

Stomatological disease such as ulcers, edema, exudation in the oropharyngeal mucosa before radiotherapy

Women who are pregnant or breastfeeding

Patients allergic or sensitive to any of the compounds in the gel or study medications

Presence of lesions that completely occlude the upper digestive tract

Patients with a history of disorders, specifically those with psychotic psychiatric disorders such as schizophrenia, schizoaffective disorder, and delusional disorder, and substance/alcohol abuse

Patients participating or who have participated in another clinical trial in the last 30 days

Another uncontrollable, severe, hemodynamically unstable concurrent medical condition requiring urgent attention or threatening the patient's life

Receiving chemotherapy regimens with delayed toxicity within the last 4 weeks (six weeks for nitrosourea or mitomycin C) or continuous or weekly chemotherapy regimen with limited potential for delayed toxicity within the last two weeks

Any evidence of oral infection or disease in the oral cavity other than HNSCC

Any important medical disease or incidental abnormal laboratory finding that could increase the participant's risk in the study (based on the investigator's judgment)

Concomitant therapy with drugs that inhibit or enhance opioid action

Hypersensitivity to opioids, respiratory depression, obstructive airway disease, acute liver disease, seizure disorder, increased intracranial pressure, paralytic ileus, patients with known sensitivity to morphine, pheochromocytoma, acute asthma exacerbations, history of cardiac arrhythmia, heart failure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of superficial bacterial and fungal infections | From the first day of TV5M01 application (initiated at diagnosis of mucositis during radiotherapy) through completion of radiotherapy (approximately 7 weeks) plus 30 days after the last radiotherapy cycle, for a total duration of approximately 10-11 week
  To assess the safety profile of TV5M01 by measuring the occurrence of oral and pharyngeal superficial bacterial and fungal infections throughout the treatment period. These infections will be diagnosed through clinical examination and confirmed by culture testing when appropriate. The comparative incidence rates between the treatment arms will be analyzed using Fisher's exact test to determine any statistically significant differences in infection risk. This endpoint is critical for evaluating the local mucosal safety of the intervention, particularly given the immunocompromised status of patients undergoing radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Valle del Lili, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No
Data publication policy: Our identifiable personal data (IPD) is not publicly available to protect participant privacy and confidentiality. We do not plan to share individual participant data with external researchers due to: 1) local regulatory restrictions, 2) the sensitive nature of the medical information collected, 3) limitations in our institutional data sharing infrastructure, and 4) commitments made to participants during the informed consent process regarding data confidentiality. Our ethics committee has approved this data management approach in accordance with Colombian regulations.

REFERENCES:
- [Background] Rosati M, Bramante S, Conti F, Frattari A, Rizzi M, Roman RA. Operative Gynecological Laparoscopy Under Conscious Sedation. JSLS. 2020 Apr-Jun;24(2):e2020.00020. doi: 10.4293/JSLS.2020.00020. PMID 32612345
- [Background] Liu YP, He RX, Chen ZH, Kang LL, Song JQ, Liu Y, Shi CY, Chen JY, Dong H, Zhang Y, Li MQ, Jin Y, Qin J, Yang YL. Case report: An asymptomatic mother with an inborn error of cobalamin metabolism (cblC) detected through high homocysteine levels during prenatal diagnosis. Front Nutr. 2023 May 12;10:1124387. doi: 10.3389/fnut.2023.1124387. eCollection 2023. PMID 37252234
- [Background] Gramegna A, Amati F, Terranova L, Sotgiu G, Tarsia P, Miglietta D, Calderazzo MA, Aliberti S, Blasi F. Neutrophil elastase in bronchiectasis. Respir Res. 2017 Dec 19;18(1):211. doi: 10.1186/s12931-017-0691-x. PMID 29258516
- [Background] Mourad R, Kolisnyk S, Baiun Y, Falk A, Yuriy T, Valerii F, Kopeev A, Suldina O, Pospelov A, Kim J, Rusakov A, Lebl DR. Performance of hybrid artificial intelligence in determining candidacy for lumbar stenosis surgery. Eur Spine J. 2022 Aug;31(8):2149-2155. doi: 10.1007/s00586-022-07307-7. Epub 2022 Jul 8. PMID 35802195
- [Background] Oit-Wiscombe I, Virag L, Soomets U, Altraja A. Increased DNA damage in progression of COPD: a response by poly(ADP-ribose) polymerase-1. PLoS One. 2013 Jul 24;8(7):e70333. doi: 10.1371/journal.pone.0070333. Print 2013. PMID 23894640
- [Background] Skeie EJ, Borge JA, Leboeuf-Yde C, Bolton J, Wedderkopp N. Reliability of diagnostic ultrasound in measuring the multifidus muscle. Chiropr Man Therap. 2015 Apr 15;23:15. doi: 10.1186/s12998-015-0059-6. eCollection 2015. PMID 25878771
- [Background] Cerchietti LC, Navigante AH, Bonomi MR, Zaderajko MA, Menendez PR, Pogany CE, Roth BM. Effect of topical morphine for mucositis-associated pain following concomitant chemoradiotherapy for head and neck carcinoma. Cancer. 2002 Nov 15;95(10):2230-6. doi: 10.1002/cncr.10938. PMID 12412178
- [Background] Zhu W, Mei H, Jia L, Zhao H, Li X, Meng X, Zhao X, Xing L, Yu J. Epigallocatechin-3-gallate mouthwash protects mucosa from radiation-induced mucositis in head and neck cancer patients: a prospective, non-randomised, phase 1 trial. Invest New Drugs. 2020 Aug;38(4):1129-1136. doi: 10.1007/s10637-019-00871-8. Epub 2019 Nov 7. PMID 31701429